CLINICAL TRIAL: NCT03799042
Title: The Use of Virtual Reality (VR) and the Change in Emotional State in Hong Kong Elders
Brief Title: The Use of Virtual Reality (VR) and the Change in Emotion in Hong Kong Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kelvin KF Tsoi, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CUHKHKT0818
Record Dates: First submitted 2018-08-10; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Virtual Reality; Emotions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitural Reality (Experimental): Virtual Reality 3D glass
  Interventions: Device: Virtual Reality
- Inter-generation interaction (Active Comparator): Elders-teenager interaction
  Interventions: Behavioral: Inter-generation interaction

INTERVENTIONS:
Device: Virtual Reality — Subjects will wear a 3D glass and watch 3D pictures (or video) of landscapes or tourist sites in Hong Kong.
  Arms: Vitural Reality
Behavioral: Inter-generation interaction — Secondary school student will play games and chats with secondary school students. Games involve identifying famous landscapes or tourist sites in Hong Kong
  Arms: Inter-generation interaction

SUMMARY:
Virtual Reality (VR) is a technology that combines virtual technology and real-world scenario. In recent years, more and more neuroscience and psychology scientists utilised VR technology in their research. In Hong Kong, many of the community-dwelling elders are immobile. Long-term homestay may negatively affect the emotional state. Measuring the emotional change after administration of VR may prove it as an alternative tool for emotion intervention.

The primary objective is to compare the improvement in the emotional changes between intergeneration interaction and the use of VR technology.

The secondary objective is to evaluate the side effect after using VR technology.

This is a randomized, open label-controlled trial with a crossover design. The subject will be randomized in a ratio of 1:1 into two different intervention groups, the VR group and the Intergeneration Interaction group. After 2 weeks of washout period, the VR group will receive Intergeneration Interaction and vice versa. The intervention phases last approximately 2 hours. The change in the emotional state will be assessed using the Positive and Negative Affect Scale. Any adverse event that causes by the VR will be recorded using the Simulator Sickness Questionnaire(SSQ).

This trial is the first study in Hong Kong to investigate the change of emotional state after the administration of VR technology, targeting community-dwelling elders in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Native Cantonese Speaker

Exclusion Criteria:

-

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | Major assessment points are scheduled prior to intervention(baseline), post intervention of the first visit (approximate 2 hours after baseline), and post intervention of the second visit (2 weeks after first intervention.)
  Measure the difference in mean score between the two intervention groups. The Positive and Negative Affect Schedule (PANAS) is consist of 20 emotions. Positive Affect Score consists of 10 positive emotions, while Negative Affect Score consists of 10 negative emotions. Positive Affect Score ranges from 10 to 50, a score of 30 indicates a higher level of positive emotion. Negative Affect Score ranges from 10 to 50, a score of 15 indicates a higher level of negative emotion. Total PANAS score is 100, added up by both Positive Affect Score and Negative Affect Score.

SECONDARY OUTCOMES:
Simulator Sickness Questionnaire | Major assessment points are scheduled prior to intervention(baseline), post intervention of the first visit (approximate 2 hours after baseline), and post intervention of the second visit (2 weeks after first intervention.)
  Measure the difference in mean score between the two intervention groups. The Simulator Sickness Questionnaire (SSQ) is consist of 16 symptoms. Each symptom includes four level, none (0 marks), slight(1mark), moderate (2 marks) and severe(3). Three subscore are included, Nausea-related subscore (Symptom 1,6,7,8,9,15,16), Oculomotor-related subscore (Symptom 1,2,3,4,5,9,11), and Disorientation-related subscore (5,8,10,11,12,13,14). Adding Nausea subscore, oculomotor subscore, and disorientation subscore and multiply by 3.74. Total score larger than 15 indicated a significant level of adverse reaction.
Positive and Negative Affect Schedule (PANAS) | Major assessment points are scheduled prior, post-intervention of first visit (approximate two hours after baseline)
  Measure the changes from baseline to first intervention
Simulator Sickness Questionnaire | Major assessment points are scheduled prior, post-intervention of first visit (approximate two hours after baseline)
  Measure the changes from baseline to first intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin KF Tsoi, BSc, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Caritas Elderly Centre - Sai Kung, Hong Kong, HK, Hong Kong